CLINICAL TRIAL: NCT02767154
Title: A Randomized Controlled Trial Comparing Dextran-based Priming (PrimECC), and Standard Crystalloid and Mannitol-based Priming Solution in Adult Cardiac Surgery
Brief Title: Dextran-based Priming vs. Crystalloid and Mannitol-based Priming Solution in Adult Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Anders Jeppssons, MD, PhD, Professor/Senior consultant, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1003-15
Record Dates: First submitted 2016-04-12; First posted 2016-05-10 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Heart Disease
Keywords: extracorporeal circulation
MeSH Terms: conditions — Heart Diseases | interventions — Extracorporeal Circulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PrimECC (Active Comparator): 1250 ml of a priming solution based on the colloid Dextran 40 to use for extracorporeal circulation.
  Interventions: Device: A colloid Dextran 40 solution for extracorporeal circulation
- Ringer-Acetate/Mannitol (Active Comparator): 1250 ml of a priming solution based on the crystalloid Ringer-Acetate (1000ml) and Mannitol (250ml).
  Interventions: Device: Ringer-Acetate and Mannitol

INTERVENTIONS:
Device: A colloid Dextran 40 solution for extracorporeal circulation — The oncotic pressure of the PrimECC solution is higher than that of a crystalloid Ringer-acetate/mannitol solution. It should maintain the plasma oncotic pressure during and after cardiopulmonary bypass (CPB). Subsequently, the leakage of fluids from the systemic circulation to the interstitial compartment during CPB can be reduced, and a higher plasma volume and a better fluid balance can be achieved.
  Other Names: PrimECC
  Arms: PrimECC
Device: Ringer-Acetate and Mannitol — Currently clinic standard for priming the CPB circuit.
  Other Names: Standard crystalloid prime
  Arms: Ringer-Acetate/Mannitol

SUMMARY:
This study will compare two priming solutions for extracorporeal circulation, one based on Dextran 40, one based on crystalloid and mannitol. Primary endpoint is oncotic pressure during cardiopulmonary bypass. Secondary endpoints included fluid balance and organ functions.

DETAILED DESCRIPTION:
This is a prospective, single center, double-blinded, randomized controlled clinical trial. Eighty patients are randomized 1:1 to either cardiopulmonary bypass with the dextran-based solution or standard priming with Ringer-Acetate and Mannitol.

Primary endpoint will be oncotic pressure during cardio pulmonary bypass. Secondary endpoints include perioperative fluid balance, coagulation, platelet function, postoperative bleeding volume, transfusion requirements, renal function, liver function, pulmonary function, inflammatory activation and markers for brain and heart injury.

Blood samples for oncotic pressure measurements will be collected from an arterial line before and during surgery. Organ function will be assessed before surgery and 2 hours cardio pulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 - 75 years
* Elective cardiac surgery procedure with expected CBP time above 90 minutes
* Subject provides a legally effective informed consent.

Exclusion Criteria:

* Known previous cardiac surgery
* Coagulation disorder
* Malignancy
* Kidney failure
* Liver failure
* Ongoing septicaemia
* Ongoing antithrombotic treatment other than acetylsalicylic acid
* Systemic inflammatory disorders treated with corticosteroids
* Not able to understand Swedish

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-07-12 (Actual); Study Completion 2017-07-13 (Actual)

PRIMARY OUTCOMES:
Change in oncotic pressure in plasma | After 1 hour of cardiopulmonary bypass
  The oncotic pressure in plasma is measured using an Osmomat 050 and reported in kPa. Points of measurement is before ECC and at 60 minutes into ECC

SECONDARY OUTCOMES:
Change in fluid balance | Within 24 hours after cardiopulmonary bypass
  Patient fluid balance is registered from ECC-start until 24 hours post-ECC. Infusion of crystalloids and colloids and urine output is registered in ml.
Amount of bleeding | Within 24 hours after cardiopulmonary bypass
  Bleeding is registered from ECC-start until 24 hours post-ECC. Intraoperative bleeding and postoperative chest tube drainage for 24 hours are added and registered in ml.
Amount of transfusions | Within 24 hours after cardiopulmonary bypass
  Transfusions of red blood cells, platelets and plasma from ECC-start until 24 hours post-ECC are registered and reported in ml.
Change in coagulation (1). | Within 2 hours after cardiopulmonary bypass
  Blood samples will be analyzed with modified rotational thromboelastometry (ROTEM) and calibrated automated thrombography. Points of measurement will be before ECC and at 2 hours post-ECC. Results will be reported as normal, above normal or below normal.
Change in coagulation (2). | Within 2 hours after cardiopulmonary bypass
  Blood samples will be analyzed calibrated automated thrombography. Points of measurement will be before ECC and at 2 hours post-ECC. Results will be reported as normal, above normal or below normal.
Change in platelet function | Within 2 hours after cardiopulmonary bypass
  Platelet function will be measured with impedance aggregometry (Multiplate). Points of measurement will be before ECC and at 2 hours post-ECC. Results will be reported as normal or below normal.
Change in renal function (1) | Within 2 hours after cardiopulmonary bypass
  Renal function is measured as µmol/L of Creatinine in serum. Points of measurement will be before ECC and at 2 hours post-ECC.
Change in renal function (2) | After 1 hour of cardiopulmonary bypass
  Renal tubular damage is measured by analysis of U-NAG. Urine is collected before ECC and at 60 minutes into ECC. Results will be reported as U-NAG/U-Creatinine ratio (U/min).
Change in liver function (1) | Within 2 hours after cardiopulmonary bypass
  The liver function is measured as µkat/L of ASAT in serum. Points of measurement will be before ECC and at 2 hours post-ECC.
Change in liver function (2) | Within 2 hours after cardiopulmonary bypass
  The liver function is measured as µkat/L of ALAT in serum. Points of measurement will be before ECC and at 2 hours post-ECC.
Change in pulmonary function | Within 2 hours after cardiopulmonary bypass
  The pulmonary function is measured by arterial blood gases assessing PaO2/FiO2 and reported in mmHg. Points of measurement will be before ECC and at 2 hours post-ECC.
Change in ischemic heart injury marker. | Within 24 hours after cardiopulmonary bypass
  The ischemic status of the heart is measures as ng/L of highly sensitive Troponin-T. Points of measurement will be before ECC and at 24 hours post-ECC.
Change in brain injury marker (1) | Within 2 hours after cardiopulmonary bypass
  Brain damage is measured as ng/L Tau in plasma. Points of measurement will be before ECC and at 2 hours post-ECC.
Change in brain injury marker (2) | Within 2 hours after cardiopulmonary bypass
  Brain damage is measured as ng/L of NFL in serum. Points of measurement will be before ECC and at 2 hours post-ECC.
Change in brain injury marker (3) | Within 2 hours after cardiopulmonary bypass
  Brain damage is measured as µg/L of S100B in serum. Points of measurement will be before ECC and at 2 hours post-ECC.
Change in brain injury marker (4) | Within 2 hours after cardiopulmonary bypass
  Brain damage is measured as µg/L of NSE in serum. Points of measurement will be before ECC and at 2 hours post-ECC.
Change in inflammatory activation | Within 2 hours after cardiopulmonary bypass
  Inflammatory activation is measured as ng/L of IL-6 in plasma. Points of measurement will be before ECC and at 2 hours post-ECC.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, VGR, Sweden

IPD SHARING:
Plan to Share IPD: No